CLINICAL TRIAL: NCT05837936
Title: A Prospective Observational Study Evaluating Extubation Criteria in Children Less 10 Years of Age and Younger Undergoing Intravenous Anesthesia
Brief Title: Total Intravenous Anesthesia (TIVA)/Sevoflurane Initiated Intravenous Anesthesia (SIIVA) in Pediatric Patients
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00092312
Record Dates: First submitted 2023-04-03; First posted 2023-05-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Extubation
Keywords: anesthesia; Propofol; inhalational agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total intravenous anesthesia (TIVA): TIVA is achieved without inhalational agents and may be performed in cases where patients have an intravenous line in place prior to induction of anesthesia
  Interventions: Other: Total intravenous anesthesia (TIVA)
- Sevoflurane initiated intravenous anesthesia (SIIVA): SIIVA is a modification of TIVA in the setting where a patient does not tolerate the insertion of an intravenous line prior to induction of anesthesia. The patient undergoes induction of anesthesia with sevoflurane and transition to Propofol IV anesthesia for maintenance once the intravenous line is in place and discontinues the inhalational agent, sevoflurane.
  Interventions: Other: Sevoflurane initiated intravenous anesthesia (SIIVA)

INTERVENTIONS:
Other: Total intravenous anesthesia (TIVA) — TIVA anesthetic -no inhalational gases for surgery
  Groups: Total intravenous anesthesia (TIVA)
Other: Sevoflurane initiated intravenous anesthesia (SIIVA) — SIIVA - sevoflurane anesthetic gases for surgery
  Groups: Sevoflurane initiated intravenous anesthesia (SIIVA)

SUMMARY:
Because Propofol is the primary "anesthetic agent," and inhalational agents remain in trace quantities at the end of the procedure Sevoflurane initiated intravenous anesthesia (SIIVA) or not present at all Total intravenous anesthesia (TIVA) it is likely that different criteria may be predictive of extubation success in these patients compared to inhalational anesthesia.

DETAILED DESCRIPTION:
This is because these anesthetic regimens have different pharmacologic mechanisms of actions, and therefore interact with central nervous system in different ways leading to potentially the need for different extubation criteria in patients receiving TIVA or SIIVA. Additionally, intravenous agents likely have less of an effect on airway reflexes and ventilation at light levels of anesthesia. This study is proposing an observational study to examine the predictive value of various extubation criteria in the setting of SIIVA and TIVA.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients <10 years of age
* Undergoing elective or emergency surgery with planned airway instrumentation with an endotracheal tube (ETT)
* Patients having general anesthesia with a planned SIIVA or TIVA technique
* Patients with an end tidal agent concentration of Sevoflurane<0.1% at the time of emergence and extubation
* following sevoflurane induction to place IV

Exclusion Criteria:

* History of home oxygen use or ventilator dependence
* Patients with cyanotic congenital heart disease
* Patients undergoing anesthesia for imaging procedures alone
* Patients intended to be managed with supraglottic airway
* Patients having an anesthesia time < 30 minutes
* Monitored Anesthesia Care (not general anesthesia)
* Patients with contraindication to receiving Propofol (i.e. mitochondrial myopathy)

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All study participants must be < 10 years of age and undergoing general anesthesia and surgery with an endotracheal tube and using a SIIVA or TIVA approach
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Extubation success rate | Day 1
  quality of extubation will be assess using a standard rubric for all extubation

SECONDARY OUTCOMES:
Rate of extubation that requiring intervention | Day 1
  desaturation, laryngospasm, airway obstruction or other issues

OTHER OUTCOMES:
Number of Subjects that met specific extubation criteria | Day 1
  Assess the presence of specific extubation criteria met during the extubation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas "Wes" Templeton, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States
- Perth Children's Hospital, Perth, Australia

IPD SHARING:
Plan to Share IPD: Undecided